CLINICAL TRIAL: NCT03925740
Title: The Effectiveness of Casein Phosphopeptide Amorphous Calcium Phosphate (MI Varnish) and 5% Sodium Fluoride Plus Xylitol (PreviDent Varnish) on Non Cavitated Interproximal Lesions. Randomised Clinical Trial
Brief Title: MI and PreviDent Varnish on Non Cavitated Interproximal Lesions.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Narmin Helal, Assistant Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KAUFDNHelal
Record Dates: First submitted 2019-04-21; First posted 2019-04-24 (Actual); Last update posted 2020-04-09 (Actual); Status verified 2020-04

CONDITIONS: Prevention
Keywords: caries; interproximal caries; MI varnish; PreviDent varnish; Fluoride; 1.23% APF Fluoride
MeSH Terms: interventions — casein phosphopeptide-amorphous calcium phosphate nanocomplex

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- MI Varnish Group (Experimental): The teeth will be cleaned, plaque will be removed, placement of wedge/separator and teeth will be dried with the aids of light, mouth mirror and dental probe following ICDAS score. Remineralization protocol, group one will be treated with MI varnish according to the manufacture instructions in first visit and each follow up visits.
  Interventions: Drug: MI Varnish
- PreviDent Varnish Group (Experimental): The teeth will be cleaned, plaque will be removed, placement of wedge/separator and teeth will be dried with the aids of light, mouth mirror and dental probe following ICDAS score. Group two will receive PreviDent varnish according to the manufacture instructions in the first visit and each follow up visits.
  Interventions: Drug: PreviDent Varnish
- 1.23% APF Control Group (Active Comparator): Regular application of APF for 4 minutes with high volume suction to the whole mouth.
  Interventions: Drug: 1.23% APF

INTERVENTIONS:
Drug: MI Varnish — Application of MI varnish material versus the standard 1.23% APF.
  Other Names: GC MI varnish, Recaldent, primary DI number: D6580052651
  Arms: MI Varnish Group
Drug: PreviDent Varnish — Application of PreviDent Varnish material versus the standard 1.23% APF.
  Other Names: Colgate PreviDent varnish ,product DI number: 00038341330937
  Arms: PreviDent Varnish Group
Drug: 1.23% APF — Standard 1.23% APF application
  Other Names: ZAP fluoride gel, NDC Number: 24794-0102-16
  Arms: 1.23% APF Control Group

SUMMARY:
Fluoride products are proven to be cost effective in preventing dental caries. Newer Fluoride products have been released in the market with different components that may have an impact on the clinical and radiographic outcome regarding incipient caries management. The objective of the study is to compare the effectiveness of PreviDent and MI varnish to (1.23%) Acidulated phosphopeptide Fluoride (APF) on remineralisation of non-cavitated proximal incipient lesions.

DETAILED DESCRIPTION:
The patients will be randomly assigned in three groups by coin toss after obtaining the consent form and filling the questionnaire about file number, gender, socioeconomic status, education and occupation of the parents and their marital status. Group one will receive MI varnish, group two will receive PreviDent varnish, group three will receive 1.23% APF standard Fluoride application. The teeth will be cleaned, plaque will be removed, placement of wedge/separator and teeth will be dried with the aids of light, mouth mirror and dental probe followingInternational Caries Detection and Assessment System (ICDAS) score. The clinical assessment will be conduct during the application visit initial (T1), three months follow up visit (T2) six months follow up visit (T3) and twelve months follow up visit (T3) to evaluate the effectiveness of the different types of Fluoride. The radiographic assessment will be conducted during (T3) and (T4).

ELIGIBILITY:
Inclusion Criteria:

1. Patient is 7-10 mixed dentition
2. Patients with any incipient non cavitated posterior proximal caries
3. Patients with any incipient non cavitated anterior proximal cariesanterior
4. ICDAS Score 1 or 2

Exclusion Criteria:

1. Any patients with any serious chronic medical problem.
2. caries that cross the dentin-enamel junction (DEJ) or enamel discontinuity
3. history of proximal restorations
4. history of resin infiltrate
5. ICDAS score of proximal caries more than two clinically or radiographically.

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-05-29 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Radiographic outcome | 1 year
  Incipient lesions either remained the same or worsened.

SECONDARY OUTCOMES:
Clinical examination | 1 year
  Lesion cavitation

CONTACTS AND LOCATIONS:
Overall Officials: Heba J Sabbagh, PHD, Principal Investigator — King Abdulaziz University
Locations (1):
- King Adbulaziz University Dental Hospital, Jeddah, Mecca Region, Saudi Arabia